CLINICAL TRIAL: NCT02596802
Title: Pilot Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in Severe Left Congenital Diaphragmatic Hernia (CDH)
Brief Title: Fetoscopic Endoluminal Tracheal Occlusion (FETO) for Congenital Diaphragm Hernia
Acronym: FETO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony Johnson (Other)
Responsible Party: Sponsor-Investigator, Anthony Johnson, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HSC-MS-15-0796
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Fetoscopic Endoluminal Tracheal Occlusion; Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- FETO therapy (Experimental): Intervention name: FETO therapy
  Interventions: Device: FETO therapy

INTERVENTIONS:
Device: FETO therapy — Fetoscopic surgery at 27 to 31 weeks and 6 days gestation.

SUMMARY:
The goal is to assess the feasibility and safety of implementing Fetoscopic Endoluminal Tracheal Occlusion (FETO) therapy in fetuses with severe left Congenital Diaphragmatic Hernia (CDH) at UTHealth. UTHealth's success in this study (with an initial 5 patients) will determine the feasibility of UTHealth's future participation in multi-center trials of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years and older
* Singleton pregnancy
* Normal fetal karyotype with confirmation by culture results. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks
* Isolated Left CDH with liver up
* O/E LHR < 30% - Gestation age at time of enrollment prior to 29 wks plus 5 days as determined by clinical information (LMP, 1st or 2nd trimester ultrasound) and evaluation of first ultrasound (measured at 270 to 296 weeks) at the time of surgery
* Gestational age at FETO procedure with O/E LHR < 30% at 27 weeks 0 days to 29 weeks 6 days as determined by clinical information (LMP) and evaluation of first ultrasound
* Patient meets psychosocial criteria
* Informed consent

Exclusion Criteria:

* Patient < 18 years of age
* Multi-fetal pregnancy
* History of natural rubber latex allergy
* Preterm labor, cervix shortened (<15 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Psychosocial ineligibility, precluding consent: Inability to reside within 30 minutes of The Fetal Center at Children's Memorial Hermann Hospital. and inability to comply with the travel for the follow-up requirements of the trial; Patient does not have a support person (e.g. spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at The Fetal Center at Children's Memorial Hermann Hospital.
* Right sided CDH or bilateral CDH, isolated left sided with O/E LHR ≥25% (measured at 18 weeks 0 days to 29 weeks 5 days) as determined by ultrasound[1]
* Additional fetal anomaly and chromosomal abnormalities by ultrasound, MRI, or echocardiogram at the fetal treatment center. No cases will be removed post hoc if abnormalities are discovered in the course of post-operative monitoring
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accrete) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
* Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
* There is no safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Successful placement of Balt Goldbal2 balloon | 7 weeks after placement
Successful removal of Balt Goldbal2 balloon | within 5 weeks prior to delivery
Gestational age at delivery | at delivery

SECONDARY OUTCOMES:
Lung volume | 7 weeks after placement of balloon
Lung head ratio | 7 weeks after placement of balloon
Survival at 30 days | 30 days post delivery

OTHER OUTCOMES:
Maternal complications | After Insertion of Balloon to delivery- (from 27 weeks gestational age up to 39 weeks gestational age)
  Maternal complications include preterm labor, premature preterm rupture of membranes, oligohydramnios, polyhydramnios, and chorioamnionitis.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Johnson, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No